CLINICAL TRIAL: NCT04932967
Title: Use of Neutralizing Monoclonal Antibodies for the Treatment of COVID-19 in Patients With Hematological Malignancies (SIE-GIMEMA Study)
Brief Title: Use of nMoABs for the Treatment of COVID-19 in Patients With HM.
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: EMATO0321
Record Dates: First submitted 2021-06-17; First posted 2021-06-21 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Covid19; Hematological Malignancy
Keywords: Neutralizing Monoclonal Antibodies
MeSH Terms: conditions — COVID-19; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multicenter retrospective, non-interventional observational study to evaluate the efficacy of nMoAbs in HM patients.

DETAILED DESCRIPTION:
This is a multicenter retrospective, non-interventional observational study. The participating centres will retrospectively review all episodes of SARS-CoV-2 infection occurring in HMs identified at their institutions from February 2020 to May 2021 and treated with nMoAbs, to evaluate their efficacy.

ELIGIBILITY:
Inclusion Criteria:

* All patients must meet all the following criteria for study entry:

  1. Age equal to or greater than 18 years of age.
  2. Diagnosis of HM (acute leukemias, myelodysplastic syndromes, myeloproliferative neoplasms, lymphomas, myeloma, chronic myeloprolipherative disorders) at any stage/status.
  3. Third generation rapid molecular or antigen test positive for SARS-CoV-2 from February 2020 until May 2021
  4. Treatment with anti SARS CoV 2 nMoAbs approved by AIFA
  5. Not hospitalized for COVID-19 at the time of nMoAbs administration
  6. Not on oxygen therapy at the time of nMoAbs administration
  7. At least one of the following symptoms for no more than 10 days:

     * Fever
     * Cough
     * Anosmia
     * Ageusia / dysgeusia
     * Pharyngodynia
     * Asthenia
     * Headache
     * Nausea
     * Diarrhea
     * Myalgia
     * Dyspnea
     * Tachypnea
  8. Signed written informed consent according to ICH/EU/GCP and national local laws (if applicable).

Exclusion Criteria:

* 1. Hematological diseases, other than HM.

  2. Not tested positive for SARS-CoV-2

  3. Patients in disease remission "off therapy" for more than 6 months

  4. Immune plasma treatment in the previous two months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients older than 18 years of age with HM who received nMoAbs, approved by AIFA, for the treatment of SARS-CoV-2 infection.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
time to SARS-nCov-2 test negativization | 3 months
  To assess the efficacy of nMoAbs in infected HM patients compared to the historical control

CONTACTS AND LOCATIONS:
Locations (14):
- Italy (14):
  - Aou Consorziale Policlinico - Uo Ematologia Con Trapianto, Bari
  - Asst Degli Spedali Civili Di Brescia, Brescia
  - Ospedale Valduce - Uos Ematologia, Como
  - Aou Careggi, Florence
  - Irccs Aou San Martino, Genova
  - Fondazione Irccs "Istituto Nazionale Tumori", Milan
  - Aou Maggiore Della Carità Di Novara, Novara
  - AOU Padova, Padua
  - Aou Pisana - Uo Ematologia Universitaria, Pisa
  - Fondazione Policlinico Universitario Agostino Gemelli-Irccs, Roma
  - Aou "San Giovanni Di Dio E Ruggi D'Aragona" - Salerno - Uoc Ematologia E Trapianti Di Cellule Staminali Emopoietiche, Salerno
  - Aou Senese, Siena
  - Asui Di Udine, Presidio Ou "S. Maria Della Misericordia", Udine
  - Asst Dei Sette Laghi, Ospedale Di Circolo E Fondazione Macchi, Varese

REFERENCES:
- [Derived] Marasco V, Piciocchi A, Candoni A, Pagano L, Guidetti A, Musto P, Bruna R, Bocchia M, Visentin A, Turrini M, Tucci A, Pilerci S, Fianchi L, Salvini M, Galimberti S, Coviello E, Selleri C, Luppi M, Crea E, Fazi P, Passamonti F, Corradini P. Neutralizing monoclonal antibodies in haematological patients paucisymptomatic for COVID-19: The GIMEMA EMATO-0321 study. Br J Haematol. 2022 Oct;199(1):54-60. doi: 10.1111/bjh.18385. Epub 2022 Jul 30. PMID 35906881